CLINICAL TRIAL: NCT02214875
Title: Increasing Retention-in-care of HIV Positive Women in PMTCT Services Through Continuous Quality Improvement -Break Through Series in Primary & Secondary Health Care Facilities in Nigeria: A Cluster Randomized Controlled Trial
Brief Title: Lafiyan Jikin Mata "Excellent Health for Mothers"
Acronym: LJM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Integrated Health Programs, Nigeria (Other)
Collaborators: Federal Ministry of Health, Nigeria (Other Government); World Health Organization (Other); Foreign Affairs, Trade and Development, Canada (Other)
Responsible Party: Principal Investigator, DR BOLA OYELEDUN, Chief Executive Officer, Centre for Integrated Health Programs, Nigeria
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: C6-TSA-037
Record Dates: First submitted 2014-07-16; First posted 2014-08-12 (Estimated); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Retention
Keywords: Retention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CQI/BTS (Experimental): Experimental: CQI/BTS
  CQI/BTS interventions will be applied through rapid structured cycles of data collection, testing of solutions and review of changes will be done. At each site, Quality Improvement Teams (QIT) will be established among facility staff. Local Government/State QI teams will provide oversight function of facility based QI initiatives. Break Through Collaborative Series (BTS) will hold quarterly in each study state at a central location with participants from intervention sites. Sessions will provide opportunity for teams to learn from each other; adapt and implement changes using the Plan-Do-Study-Act (PDSA) model. Process indicators will be used to measure quality improvement from the intervention sites and collaboratives.
  Interventions: Other: CQI/BTS
- Control (Other): Facilities in control will continue will routine unstructured, irregular continuous quality improvement. Break Through Collaborative will not be applied to the control facilities.
  Interventions: Other: Control

INTERVENTIONS:
Other: CQI/BTS — Application of CQI/BTS interventions through employing rapid structured cycles of data collection, testing of solutions and review of changes will be implemented. At each site a Quality Improvement Team (QIT) will be established from among the facility staff. Local Government and State level QI teams will provide oversight function of the health facilities' QI initiatives. BTS as a collaborative learning approach will be conducted quarterly in each study state at a central location with participants from the intervention sites. The sessions will provide opportunity for teams to learn from each other and to adapt and implement changes using the Plan-Do-Study-Act (PDSA) model.
  Arms: CQI/BTS
Other: Control — Facilities in control will continue will routine unstructured, irregular continuous quality improvement. Break Through Collaborative will not be applied to the control facilities.
  Arms: Control

SUMMARY:
This study aims to address the research question: Will continuous quality improvement, using a Break Through Series approach, increase uptake of PMTCT services and retention-in-care of HIV-infected pregnant women and mothers at six and 12 months postpartum?

Continuous Quality Improvement (CQI) is a health systems intervention to assist programs to systematically improve services and health outcomes. The Break Through Series (BTS) is a specific CQI approach is a short-term (6- to 15-month) learning system that brings together teams from several hospitals or clinics ("collaboratives") to seek improvement in a focused topic area through a common process of data sharing and review Primary Objective To assess whether retention-in-care of HIV-infected women at six (6) months postpartum is higher at health facilities implementing CQI-BTS approaches than at health facilities not implementing CQI-BTS approaches.

Secondary Objectives

To assess whether implementation of CQI-BTS initiatives at health facilities increases:

1. Uptake of PMTCT services by HIV-infected pregnant women;
2. Retention-in-care of HIV-infected women at twelve (12) months postpartum;
3. Retention-in-care of HIV-exposed babies at six (6) and twelve (12) months of age;
4. Uptake of a pre-defined, minimum set of integrated RH/PMTCT services by HIV-infected women in health facilities.

DETAILED DESCRIPTION:
Methods/ Study design/ Population/ Interventions Study Design: A cluster randomized controlled trial in which 32 public primary and secondary health care facilities are randomized into 16 intervention and 16 control sites. The control sites will receive routine CIHP support, while the intervention sites will receive structured CQI-BTS interventions.

Study sites Based on pre-set site selection criteria, 32 sites were selected from a total of 241 eligible sites supported by the Centre for Integrated Healthcare Programs (CIHP), to provide comprehensive HIV care and treatment programs. These sites are at higher levels of standardized care compared to Government of Nigeria sites where there is minimal standardization of care. The following criteria were used to select health facilities for the study;

* Facility supports ANC/PMTCT services and has capacity to provide ART until 12-18 months post-partum
* Onsite delivery of HIV+ women by the facility
* Provision of postpartum care follow-up for HIV+ women
* ANC attendance with at least 2 HIV+ women per month for general hospitals and at least 1 per month for primary health care (PHCs)
* Availability of, at least, two trained community health extension workers
* Facilities providing PMTCT services for more than six months prior to onset of study

Study Participants:

Participants are HIV-infected pregnant women presenting at study sites for 1st booking at antenatal clinics with gestational age of 34 weeks or less, ART naive, accept ARV and agree to remain in care for at least six months post-partum.

Control and Intervention arms:

Individual pregnant women and mothers attending facilities in the control and intervention arms receive the same routine care that includes a "test and treat" protocol i.e. same day HIV testing and initiation of triple ARVs (option B) of HIV+ pregnant women. Clients eligible for lifelong ART based on CD4 count, and/or WHO staging, continue ARVs indefinitely for their own health, while those not eligible continue ARV prophylaxis according to the National guidelines. For the purpose of this study, antenatal clients are seen for their ARV drug refills until delivery according to the National ANC schedule of appointments. Postpartum, visits follow the immunization schedule i.e. 6 weeks, 10 weeks, and 14 weeks and thereafter 2 monthly until 12 months. Facilities in the control arm continue to receive routine health system support from CIHP

Intervention package:

CQI interventions employ rapid cycles of data collection, testing of solutions and review of changes will be implemented. At each site a Quality Improvement Team (QIT) will be established from among the local staff. Local Government and State level QI teams will also be set up to provide oversight function of the health facilities' QI initiatives. The BTS is a collaborative learning approach conducted quarterly in each study state at a central location with participants from the intervention sites. The sessions provide opportunity for teams to learn from each other and to adapt and implement changes using the Plan-Do-Study-Act (PDSA) model. Driver diagrams will be developed to understand the primary and secondary drivers for low retention of HIV positive mothers and formulate action plans and indicator sets to address these. Between the collaborative sessions, specific designated improvement coaches will follow up site teams at regular intervals via physical site visits and telephone calls to guide implementation of change ideas. Different site teams will also be encouraged to communicate with each other through telephone calls and cross-site visits to strengthen learning and exchange of ideas.

Sample size estimation:

Sample size was calculated using the windows programme for epidemiologists. The CQI-BTS approach tested within the study would be deemed worthwhile if there is a 20% absolute increase in retention of mothers at 6 months (e.g. expected retention rate in the control arm: 40%; expected retention rate in the control arm: 60%). First, the minimum sample size needed under individual randomization was calculated to detect the desirable difference of proportions with a level of significance set at 95% (two-sided) and at 80% power. We found that 94 mother-infant pairs would be needed in each arm under individual randomization. Second, bearing in mind that this trial will randomize the intervention package under several clusters, the sample size from a non-cluster randomized trial was inflated by an Inflation Factor (IF). The IF is calculated as follows: IF = 1 + (m - 1) ro, where m is the size of each cluster, and ro the internal variability which represents how strongly individuals within clusters are related to each other. In our case, it is difficult to estimate a priori this internal variability due to lack of primary data: it is possible that the standardized structure of the intervention tested within the trial will lead to a relatively low cluster internal variability; alternatively, because the intervention package depends on the individual capacity/will of health-care personnel, this may increase the internal variability across clusters. Hence, we believe it is reasonable to assume a ro value of 0.10, as recommended by most authors. We set the size of cluster at 20, which gave an inflation factor of 2.9. Additionally, since this research is being carried out in an operational context, we allowed for up to 20% of routine data to be incomplete or maternal mortality in pregnancy and therefore data on retention in care not available for analysis. As a conclusion, a total of 327 mother-infant pairs are needed in each arm. There will be 16 clusters in each arm with a minimum number of 20 HIV-infected pregnant women per site. A total of 640 pregnant HIV-infected women will be recruited.

Data management plan:

Primary outcome data is sourced from the local health registers -Data collection and entry occur weekly in both study arms by research assistants. A monthly review of these data is conducted by the LJM study team. In addition, process measures are routinely collected to assess the integrity of implementation of the CQI-BTS intervention.

Primary Outcome: Proportion of HIV+ pregnant women in care 6 months postpartum Source Document: PMTCT ARV register

Secondary Outcome 1: Proportion of HIV+ pregnant women initiating ARV prophylaxis or treatment within 2 weeks of enrolment Source Document: PMTCT HCT register, PMTCT ARV register and Mother Child Care Form

Secondary Outcome 2: Proportion of HIV+ pregnant women care 12 months postpartum Source Document: PMTCT ARV register, Mother and Child Care Form

Secondary Outcome 3: Proportion of HIV exposed infants with Dry Blood Spot (DBS) samples taken at 8 weeks of life Source Document: Child follow up register and Mother Child Care Form

Analysis plan:

Descriptive analyses will be conducted to outline participants' and clusters' baseline characteristics and outcomes by study arms using frequency tabulations and summary statistics. Bi-variate analysis will be done to identify potential prognostic factors confounding the distribution of baseline characteristics among the arms that require adjustment.

ELIGIBILITY:
Inclusion Criteria:

1. They must be pregnant women newly diagnosed for HIV during ANC
2. Clients must present with gestational age of 34weeks or less at ANC enrollment
3. They must accept in principle to take ARVs and remain in care.
4. They must be willing to participate until at least six months postpartum
5. Must be domiciled in the facility coverage area.
6. Previously diagnosed HIV positive pregnant women yet to start ART

Exclusion Criteria:

1. Clients requesting fee/remuneration for participation
2. Positive women already on ART.
3. Unbooked HIV positive pregnant woman coming in labour.
4. Positive pregnant women with gestational age more than 34 weeks.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 491 (Actual)
Dates: Start 2014-07-14 (Actual); Primary Completion 2016-10-31 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Proportion of HIV+ pregnant women in care 6 months postpartum | Six months post partum
  Denominator= Total number of HIV + pregnant women enrolled to participate in the study Numerator= Total number of HIV + pregnant women retained at six months postpartum

SECONDARY OUTCOMES:
Proportion of HIV exposed infants with Dry Blood Spot (DBS) samples taken at 6-8 months of life | 2 months post delivery of exposed infant
  Denominator: Number of HIV exposed infants delivered at facility
  Numerator: Number of exposed infants whose DBS was taken at 6-8 months of life

CONTACTS AND LOCATIONS:
Overall Officials: Bolanle Oyeledun, MASTERS, Principal Investigator — Center for Integrated Health Program(CIHP)
Locations (1):
- Center for Integrated Health Program, Abuja, Federal Capital Territory, Nigeria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Osibo B, Oronsaye F, Alo OD, Phillips A, Becquet R, Shaffer N, Ogirima F, Imarhiagbe C, Ameh B, Ezebuka O, Sodzi-Tettey S, Obi A, Afolabi OT, Inedu A, Anyaike C, Oyeledun B. Using Small Tests of Change to Improve PMTCT Services in Northern Nigeria: Experiences From Implementation of a Continuous Quality Improvement and Breakthrough Series Program. J Acquir Immune Defic Syndr. 2017 Jun 1;75 Suppl 2:S165-S172. doi: 10.1097/QAI.0000000000001369. PMID 28498186